CLINICAL TRIAL: NCT05816850
Title: Multilayer Biological Characterization of Advanced Follicular Lymphoma: a Translational Study From FIL_FOLL12 Trial
Acronym: FIL_FOLL-BIO
Status: Recruiting | Type: Observational
Sponsor: Fondazione Italiana Linfomi - ETS (Other)
Responsible Party: Sponsor
Other Study IDs: FIL_FOLL-BIO
Record Dates: First submitted 2023-04-04; First posted 2023-04-18 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-09

CONDITIONS: Follicular Lymphoma
Keywords: Lymphoma; Follicular; Immunochemotherapy; FL; Aberration; Mutation; EZH2; CHOP; Bendamustine; Biological; Rituximab; Biomarker
MeSH Terms: conditions — Lymphoma, Follicular; Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — 1. Peripheral blood and bone marrow aspirate samples previously collected from patient enrolled in FIL_FOLL12 trial
  2. Formalin-fixed paraffin-embedded samples collected from initial diagnosis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients enrolled: Patient affected by advanced Follicular Lymphoma treated with immunochemotherapy in the FIL_FOLL12 trial
  Interventions: Diagnostic Test: EZH2 mutations/CNAs by droplet digital PCR (ddPCR); Diagnostic Test: EZH2-derived gene expression signature by RNA-Seq

INTERVENTIONS:
Diagnostic Test: EZH2 mutations/CNAs by droplet digital PCR (ddPCR) — Test of EZH2 mutations/CNAs by droplet digital PCR (ddPCR) in peripheral blood and in unsorted bone marrow aspirate samples at enrolment
Diagnostic Test: EZH2-derived gene expression signature by RNA-Seq — Test of EZH2-derived gene expression signature by RNA-Seq in a subset of diagnostic FFPE samples

SUMMARY:
This is a Multicenter, Retrospective, Biological study ancillary to FOLL12 trial to evaluate the role of EZH2 aberrations in patient with FL treated with immunochemotherapy. Moreover, several novel biomarkers of FL will be investigated.

DETAILED DESCRIPTION:
Current standard first-line treatment for advanced follicular lymphoma (FL) is still represented by chemoimmunotherapy combinations, with CHOP/CVP or bendamustine (B) as the main regimens with no standard criteria to prefer one over another.

EZH2 mutations have been associated with longer progression-free survival (PFS) in patients treated with CHOP/CVP regimens, but not with Bendamustine (independently from the type of anti-CD20 therapy received).

The FIL_FOLL12 trial (NCT02063685), a large phase III trial (with a pre-planned biological material sampling) enrolling 807 advanced FL patients treated with front-line R-CHOP or bendamustine-rituximab (BR), appears an ideal platform to validate the predictive value of EZH2 and its applicability to the clinical practice.

The aim of this study is to provide to clinicians a useful and practical biomarker to guide the choice of the most effective chemotherapy backbone (in addition to anti-CD20 immunotherapy) for first line treatment of patients with advanced FL (e.g. R-CHOP for EZH2 aberrated vs BR for EZH2 wild type patients).

Moreover, to implement an Italian network of laboratories able to provide these translational outputs within a rapid turnaround time.

Finally, taking advantage of the already collected BM and PB samples, several novel biomarkers of FL heterogeneity will be investigated, in particular: EZH2 protein expression in tumor samples, alternative molecular markers for minimal residual disease (MRD), clonal hematopoiesis of indeterminate potential (CHIP), pharmacogenomics and constitutional genomics as well as microbiome profiles.

ELIGIBILITY:
Inclusion Criteria:

* Patient enrolled in the FIL_FOLL12 trial (documented by the signature of the study informed consent);
* Availability of biological samples: bone marrow aspirate, peripheral blood and/or FFPE diagnostic sample (nodal or extranodal);

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient affected by advanced Follicular Lymphoma treated with immunochemotherapy in the FIL_FOLL12 trial
Sampling Method: Non-Probability Sample
Enrollment: 654 (Estimated)
Dates: Start 2023-09-19 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | From treatment start up to 43 months
  Time between the treatment start and the first documentation of recurrence, progression or death from any cause

SECONDARY OUTCOMES:
Response rate | From treatment start to 7 months (R-Bendamustine) or from treatment start to 5,6 months (R-CHOP)
  Response rate (complete metabolic response/minimal residual disease (MRD) negativity) at the end of induction.
Concordance between EZH2 gene mutations/gains and EZH2-related gene expression signature | Before treatment start
  Concordance between EZH2 gene mutations/gains and EZH2-related gene expression signature

CONTACTS AND LOCATIONS:
Overall Officials: Simone Ferrero, MD, Principal Investigator — SC Ematologia U - AOU Città della Salute e della Scienza di Torino
Locations (26):
- Italy (26):
  - A.O. SS. Antonio e Biagio e Cesare Arrigo, S.C. Ematologia, Alessandria
  - Nuovo Ospedale degli Infermi, SSD Ematologia, Biella
  - ASST Spedali Civili di Brescia - Ematologia, Brescia
  - Azienda Ospedaliera Universitaria Policlinico - S. Marco, UOC di Ematologia, Catania
  - A.O. S. Croce e Carle, S.C. di Ematologia e Trapianto di Midollo Osseo, Cuneo
  - Azienda Ospedaliera Universitaria Careggi - Unità funzionale di Ematologia, Florence
  - Ospedale Policlinico San Martino S.S.R.L. - IRCCS per l'Oncologia, Ematologia e terapie cellulari, Genova
  - IRCCS Istituto Romagnolo per lo studio dei Tumori "Dino Amadori" - IRST S.R.L., Ematologia, Meldola
  - ASST Grande Ospedale Metropolitano Niguarda, SC Ematologia, Milan
  - Fondazione IRCCS Istituto Nazionale dei Tumori di Milano, Ematologia, Milan
  - Azienda Ospedaliero-Universitaria Policlinico di Modena, U.O. Oncologia, Modena
  - Fondazione IRCCS San Gerardo dei Tintori - Ematologia, Monza
  - AOU Maggiore della Carità di Novara, SCDU Ematologia, Novara
  - Presidio ospedaliero "A. Tortora", U.O. Onco-ematologia, Pagani
  - A.O. Ospedali Riuniti Villa Sofia-Cervello, Divisione di Ematologia, Palermo
  - IRCCS Policlinico S. Matteo di Pavia, Divisione di Ematologia, Pavia
  - Ospedale Guglielmo da Saliceto, U.O. Ematologia, Piacenza
  - Grande Ospedale Metropolitano Bianchi Melacrino Morelli - Ematologia, Reggio Calabria
  - Ospedale degli Infermi di Rimini, U.O. di Ematologia, Rimini
  - Policlinico Umberto I - Università "La Sapienza", Istituto Ematologia -Dipartimento di Medicina Traslazionale e di Precisione, Roma
  - Istituto Clinico Humanitas, U.O. Ematologia, Rozzano
  - A.O.U. Città della Salute e della Scienza di Torino, Ematologia Universitaria, Torino
  - A.O.U. Città della Salute e della Scienza di Torino, S.C. Ematologia, Torino
  - A.O. C. Panico, U.O.C Ematologia e Trapianto, Tricase
  - Azienda Sanitaria Universitaria Friuli Centrale (ASU FC), SOC Clinica Ematologica, Udine
  - Ospedale di Circolo - U.O.C Ematologia, Varese

IPD SHARING:
Plan to Share IPD: Undecided